CLINICAL TRIAL: NCT02155257
Title: A Feasibility Study: Understanding and Altering Pain Expectations in Subjects With Osteoarthritis of the Knee or Hip
Brief Title: Pain Expectations in Subjects With Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00028525
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee pain; Hip pain; Total Knee Replacement Surgery
MeSH Terms: conditions — Osteoarthritis | interventions — Modafinil; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Modafinil (Active Comparator): Modafinil 200 mg will be administered orally one time
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): A placebo will be administered orally one time
  Interventions: Drug: Placebo
- Gabapentin (Active Comparator): Gabapentin 900 mg will be administered orally one time
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Modafinil
  Other Names: Provigil
  Arms: Modafinil
Drug: Gabapentin
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test whether or not researchers can alter or change expectations on pain. The researchers will test whether there is an effect on the size of the pupil and responses to thermal heat temperatures in subjects with osteoarthritis of the knee or hip or healthy subjects for comparison.

One of 3 possible treatment groups will be administered to qualifying subjects: (1) gabapentin, a medication that is commonly used to treat nerve pain, (2) modafinil, a medication that is commonly used to treat people with narcolepsy (a disorder that causes people to fall asleep) and (3) a placebo, which is an inactive substance, like a sugar pill, that is not thought to have any effect on your disease or condition

DETAILED DESCRIPTION:
Purpose and rationale for this study: Both chronic pain and disability after total knee replacement surgery are predicted by negative cognitive-affective state, characterized by depression, anxiety, and a cognitive style dominated by catastrophizing. How this negative state results in chronic pain and disability is not known, but we hypothesize that it causes dysfunction of the release of the neurotransmitter, norepinephrine in several regions of the brain, mid-brain, and spinal cord that are important to many processes involved in recovery from surgery.

Objectives: (1) Gabapentin and modafinil will increase resting pupil diameter with a moderate effect size in patients with osteoarthritis; (2) Expectations will modify pain experience with a moderate effect size in these patients

Methods: 30 subjects with moderate average daily pain from osteoarthritis of the knee or hip or healthy subjects will be recruited and will come to the clinical research unit at Wake Forest. Informed consent will be confirmed and they will complete the questionnaires. We will take a verbal medical and medication history and obtain blood pressure and heart rate measurements. Verbal pain intensity report (0-10 from no pain to worst pain imaginable) will be obtained from a 5 second heat stimuli, separated by 30 seconds, delivered to a nonpainful area of skin on the arm as described in preliminary data. During pain testing, study subjects will sit in a comfortable chair in a low-ambient light room with their head positioned on a chin rest for continuous recording of pupil diameter using a near infrared recording system as described in preliminary data. Pupil diameter and probe temperature will be passed through an analog to digital converter and acquired at 60 Hertz (Hz) for subsequent analysis.

Five sequences of test stimuli will be presented, with a brief break in between each sequence. The first sequence will consist of 7 stimuli, from 39⁰ to 51⁰ Celsius (C) in 2⁰C increments, in ascending order. Data from this training sequence will not be used for analysis. Sequences 2 and 3 will consist of 5, 5-second stimuli, presented in random order, to generate moderate (50⁰C) and mild (47⁰C) pain (random condition). Sequences 4 and 5 will also consist of random presentation of 5 stimuli at these temperatures, but with different auditory tones 6 s prior to stimulus onset to correctly cue the stimulus temperature (cued condition).

Subjects will then be randomized to receive oral gabapentin, 900 milligram (mg), modafinil, 200 mg, or placebo, followed 2 hours later by pain testing with pupillometry, consisting of different sequences. The random and cued paradigms will be presented twice each followed by a sequence with one miscue in the positive expectation for pain direction (signal for 50⁰C but deliver 47⁰C) and one in the negative expectation for pain direction. Subjects will provide verbal pain intensity scores after each stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee or hip
* Adult (ages 18-80)
* Moderate pain (verbal score of ≥ 4 ≤ 7 on 0-10 scale for average pain intensity with normal activity)
* American Society of Anesthesiologists physical status 1-3
* Healthy subjects without pain

Exclusion Criteria:

* Pregnancy;
* Currently taking gabapentin
* Currently taking a narcotic prescription medication that is > 50 mg morphine equivalents/day
* Advanced or unstable cardiac, pulmonary, renal or hepatic dysfunction
* History of previous eye surgery
* Psychotic disorder or a recent psychiatric hospitalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Modafinil: Modafinil 200 mg will be administered orally one time
  Modafinil
- Placebo: A placebo will be administered orally one time
  Placebo
- Gabapentin: Gabapentin 900 mg will be administered orally one time
  Gabapentin
Period: Overall Study
Arm/Group | Modafinil | Placebo | Gabapentin
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Gabapentin | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 6 | 17
  Male | 6 | 3 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 10 | 9 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Resting Pupil Diameter
Description: Resting pupil diameter will be measured using an infrared camera to obtain baseline measurements 2 hours after dosing subject pupil diameter measurements will be repeated
Time Frame: Baseline and 2 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Modafinil | Placebo | Gabapentin
Number analyzed (Participants) | 10 | 10 | 10
mm
  Baseline | 64 (11.5) | 72 (12.6) | 69 (12.7)
  2 Hours | 66.9 (11.9) | 70.9 (14.5) | 66.1 (13.5)
Statistical Analysis 1: Comparison: Modafinil vs Placebo vs Gabapentin; Interaction between resting pupil diameter and correlation of cognitive-affective style to pain reporting. Note that this analysis is an INTERACTION between the primary outcome of this measure (pupil diameter) to that of the primary outcome measure of cognitive-affective style; Test type: Other; p = 0.540, Regression, Linear; Slope = .19, 95% CI 2-sided [-.39 to .76]

2. Primary Outcome: Pain Intensity Rating
Description: Pain is reported verbally after each stimulus by the subject on a scale of 0 (no pain) to 10 (worst imagineable pain). For each individual the value used is the average of all presentations of the 50 degree stimulus.
Time Frame: Reported 5 seconds after each stimulus
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil | Placebo | Gabapentin
Number analyzed (Participants) | 10 | 10 | 10
units on a scale | 3.2 (1.7) | 2.8 (1.8) | 2.8 (2.0)

3. Primary Outcome: Cognitive Style
Description: Cognitive style determined for each individual by subtracting the score in the Pain Catastrophizing Scale (CATS) questionnaire (with a score range of 0-52 with higher score showing more catastrophizing) from the Life Orientation Test Revised (LOT-R) questionnaire (score range of 0-24, with a higher score denoting a better outcome). Thus, the total score could range from ranges from -52 to 24, with lower scores indicating worse cognitive style related to pain reporting and higher scores indicating better cognitive style related to pain reporting. There are no subscales here.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modafinil | Placebo | Gabapentin
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 18.2 (2.3) | 15.5 (2.3) | 14.8 (5.7)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Modafinil | Placebo | Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-11-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT02155257/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02155257/SAP_001.pdf